CLINICAL TRIAL: NCT07349251
Title: Normal Hemostasis Values in Premature Infants
Acronym: PRHEMO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9948
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Premature Infant, Hemostasis
Keywords: Premature Infant; Neonatal Prematurity; Preterm Infants; Hemostasis
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to retrospectively determine, in a large cohort of apparently healthy children born before 37 weeks of gestation, the expected values of certain hemostasis parameters from birth to 18 months (when they start walking), and to determine whether or not they differ from those of full-term infants.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 months or younger for whom a sample was sent to the Hematology Laboratory at Strasbourg University Hospital for measurement of a hemostasis parameter

Exclusion Criteria:

* Patients with incomplete data
* Patients with a congenital hemostasis disorder (hemophilia A or B, von Willebrand disease), a coagulopathy, or hepatocellular insufficiency

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 18 months or younger for whom a sample was sent to the Hematology Laboratory at Strasbourg University Hospital for measurement of a hemostasis parameter
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11-24 (Estimated)

PRIMARY OUTCOMES:
Normal hemostasis values in premature infants | Up to 6 years
  Normal hemostasis values in premature infants will be determined according to the gestational age at birth

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Hématologie - CHU de Strasbourg - France, Strasbourg, France